CLINICAL TRIAL: NCT04605250
Title: Respiratory Variability for Respiratory Monitoring During the Postoperative Recovery Period
Acronym: VariaRessPi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19_RIPH2-01
Record Dates: First submitted 2020-07-28; First posted 2020-10-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pulmonary Complications
MeSH Terms: interventions — Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults undergoing abdominal surgery with laparotomy (Other): Respiratory variability before and after abdominal surgery
  Interventions: Other: Respiratory variability before and after surgery

INTERVENTIONS:
Other: Respiratory variability before and after surgery — The procedure consist of measuring thoracic chest movement and then calculating the respiratory variability reflected by the coefficient of variation in patients undergoing a surgery. A first recording is done during preoxygenation period using as baseline for further comparisons. (T0, 10 min) The second recording is after extubation during the postoperative recovering period, 30 minutes after interruption of sedations. (T1, 20 min, SSPI ou SIPO) The third recording is before transferring back to classical hospitalization, 1h after T1 (20 min). A fourth recording will be realized 24h after surgery for patients hospitalized in the post operative intensive care unit (T3, 20 min) Optional recordings may be realized if the patient is developing a postoperative respiratory complication during his hospital stay. A follow up for maximum 7 days consisting in consulting the medical file will be realized.

SUMMARY:
The research consist of measuring respiratory variability of several variables of the respiratory pattern at rest and during exercise using a thoracic movement measuring technique. The objective is to confirm the ability of this technique to measure the respiratory variability in healthy subjects comparing to flow measurements by a pneumotachograph. In a second step, the thoracic movement technique is applied to measure respiratory variability before and after surgery in patients after abdominal surgery with laparotomy. The objective is to observe a decrease of variability in subjects developing or at risk to develop a postoperative pulmonary complication.

DETAILED DESCRIPTION:
The incidence of Postoperative Pulmonary Complications after non-thoracic surgery varie between 2 and 19%. Postoperative Pulmonary Complications are associated with an increase of morbi-mortality and longer hospital stays. However, few possibilities are available to identify Postoperative Pulmonary Complications except predictions scores and SpO2, which decreases only face to a significant lung disease. Besides, the respiratory variability decreases during pulmonary stress situations, and is associated with an increase of mortality during mechanical ventilation. The hypothesis is that a decrease of the respiratory variability between the preoperative and the postoperative measures is associated with an increase of Postoperative Pulmonary Complications . However there is no mesuring tool of easy access in clinical practice. That is why, in a first step, a thoracic sensor belt will be tested on healthy subjects. This sensor belt is available to measure the respiratory variability.

ELIGIBILITY:
Inclusion Criteria:

* Physiological step :
* adults without any acute or chronic disease with a significant impact on daily life, particularly no cardio-respiratory disease.
* Smokers can be included.
* Free and informed consent signed.
* Clinical step :
* adults undergoing abdominal surgery with laparotomy, in emergency or scheduled,
* in Martinique and Guadeloupe.
* Free and informed oral consent.

Exclusion Criteria

* Pregnant,breast feeding women,
* minor,
* intubated patients or with criteria of imminent intubation
* subject unable to give his free and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Variation of the Tidal volume (Vt) between the preoperative and the postoperative period | 7 days
  Measure the respiratory variability in patients with abdominal surgery with laparotomy just before the anaesthetic induction and in the postoperative stage after extubation with a belt equipped with an external sensor.

CONTACTS AND LOCATIONS:
Overall Officials: BEN HASSEN Kais, MD, Principal Investigator — CHU de Martinique
Locations (1):
- CHU Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No